CLINICAL TRIAL: NCT02793102
Title: Prospective Evaluation of a Year of Therapeutic Impact Sensory Workshops on Body Mass Index in Anorexia Adolescent Mental
Brief Title: Sensory Workshops and Anorexia Nervosa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient responding to criteria
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 14-HPNCL-11
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Anorexia
Keywords: mental anorexia; sensory workshops; BMI
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olfactory workshop + Somesthesia workshop (Experimental): Olfactory workshop, Twenty odorants. Somesthesia workshop, time for moving the body, Talk Time
  Interventions: Other: Olfactory workshop; Other: Somesthesia workshop
- Auditory workshop + Somesthesia workshop (Experimental): Auditory workshop, Twenty extracts of music tracks. Somesthesia workshop, time for moving the body, Talk Time
  Interventions: Other: Somesthesia workshop; Other: Auditory workshop

INTERVENTIONS:
Other: Olfactory workshop — Twenty odorants are selected: 10 evoke a food (including 5 pleasant and unpleasant 5) and 10 suggest a non-food source
  Arms: Olfactory workshop + Somesthesia workshop
Other: Somesthesia workshop — Kinesthetic time or time for moving the body (30 min), and kinesthetic sensations (duration 10 min), and Talk Time
Other: Auditory workshop — Twenty extracts of music tracks (30 seconds each) are built in the same fashion as those used during the workshops, but are different.
  Arms: Auditory workshop + Somesthesia workshop

SUMMARY:
In the literature the use of olfactory dimension in the treatment of anorexia has not been verified experimentally. The investigator hypothesize that the therapeutic use of a dietary nature olfactory stimuli in anorexia nervosa promotes food recovery. The team propose a prospective study over a period of 12 months in which we use the Body Mass Index (BMI) as the primary endpoint of the state of anorexia nervosa patients.

DETAILED DESCRIPTION:
As part of the unit that specializes in eating disorders in adolescents, we see patients decreased taste and smell sensory abilities. Since 2006, we have implemented various sensory workshops: olfactory, tactile-kinesthetic and auditory. The establishment of this therapeutic practice that is centered on oral sphere and all respect, it was observed a decrease of 30% of the length of hospitalization. All the data we currently have in the field, suggests a rehabituation food odors and facilitate the recall of memories related to food in anorexic patients. However in the literature the use of olfactory dimension in the treatment of anorexia has not been verified experimentally. The investigator hypothesize that the therapeutic use of a dietary nature olfactory stimuli in anorexia nervosa promotes food recovery. The team propose a prospective study over a period of 12 months in which we use the Body Mass Index (BMI) as the primary endpoint of the state of anorexia nervosa patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anorexia nervosa according to DMS IV-TR (Diagnostic and Statistical Manual of Mental Disorders) criteria.
* Follow Outpatient care or hospitalization
* Able to respond to the clinical evaluation questionnaires
* Affiliated to the social security system
* Consentement Informed of the legal representative and the patient

Exclusion Criteria:

* Somatic comorbidity associated diabetes, celiac disease, brain tumor.
* Intolerance Odors, predisposition to develop asthma and / or respiratory allergies.
* Pathologie Chronic of nose and sinus.
* Hyposmic Or anosmic.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assess the impact of sensory workshops on BMI Body Mass Indexat 6 months and 12 months | Comparaison to baseline and 6 month after and maintenance at month 12
  The primary endpoint is the M6 and increase maintenance M12 BMI Body Mass Index to <or = 2.6kg / m2

CONTACTS AND LOCATIONS:
Overall Officials: Florence ASKENAZY, MD, Principal Investigator — Fondation Lenval

IPD SHARING:
Plan to Share IPD: No